CLINICAL TRIAL: NCT04628299
Title: Effects of the Myofascial Induction Technique Versus a Control Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2111201814518 B
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Foot Diseases; Myofascial Pain
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Laser (Placebo Comparator): A non-emission laser will be applied in plantar fascia
  Interventions: Other: Sham Laser
- Experimental group Myofascial Induction (Experimental): Myofascial Induction in plantar fascia
  Interventions: Other: Myofascial Induction

INTERVENTIONS:
Other: Sham Laser — Sham Laser in plantar fascia
  Arms: Sham Laser
Other: Myofascial Induction — Myofascial Induction in plantar fascia
  Arms: Experimental group Myofascial Induction

SUMMARY:
The objective is to determine the effectiveness of myofascial Induction effects on plantar pressures variables. Forty healthy subjects will be recruited for a simple blind clinical trial. All subjects will be randomly distributed in two different groups: control group (sham Laser) and experimental group (myofascial Induction). Outcome measurements will be foot plantar pressure area (footprint) by a validated platform. Two trials will be recorded before and after intervention in standing position.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without pain.

Exclusion Criteria:

* Previous lower extremities surgery
* History of lower extremities injury with residual symptoms within the last year
* Evidence of a leg-length discrepancy of more than 1 cm
* Evidence of balance deficits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Plantar pressure measure | Register a plantar pressures of foot print in standing position of 30 seconds
  Plantar pressure measure by validated footprint platform in grams / square centimeter

SECONDARY OUTCOMES:
Plantar surface measure | Register a plantar surface area of foot print in standing position of 30 seconds
  Area of plantar footprint measure by aa validated footprint platform in square centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- [Derived] Martinez-Jimenez EM, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Rodriguez-Sanz D, Trevisson-Redondo B, Romero-Morales C, Painceira-Villar R, Palomo-Lopez P, Calvo-Lobo C, Corral-Liria I. Myofascial induction technique changes plantar pressures variables compared to a simulated laser. A randomized clinical trial. J Bodyw Mov Ther. 2025 Jun;42:703-709. doi: 10.1016/j.jbmt.2025.01.029. Epub 2025 Jan 22. PMID 40325743